CLINICAL TRIAL: NCT05838963
Title: Predictive Value of Baseline CTQ-SSS Scores for Progression to Carpal Tunnel Release Surgery: A Prospective Cohort Study
Brief Title: Predictive Value of Baseline CTQ-SSS Scores for Progression to Carpal Tunnel Release Surgery: A Cohort Study
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Ahram Canadian University (Other)
Responsible Party: Principal Investigator, Mohamed Magdy ElMeligie, Lecturer of Physical Therapy and Director of Electromyography Lab, Ahram Canadian University
Other Study IDs: 012/0023444
Record Dates: First submitted 2023-04-20; First posted 2023-05-03 (Actual); Last update posted 2023-07-06 (Actual); Status verified 2023-07

CONDITIONS: Carpal Tunnel Syndrome
MeSH Terms: conditions — Carpal Tunnel Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Study Participants: This group will consist of at least 200 patients with carpal tunnel syndrome who are undergoing nonsurgical management. Participants will complete the CTQ-SSS and other functional measures at baseline, 3 months, 6 months, and 12 months. The primary outcome will be progression to carpal tunnel release (CTR) surgery. Logistic regression models will be used to assess the predictive value of baseline CTQ-SSS scores for progression to CTR surgery, adjusting for potential confounding factors such as age, sex, and baseline symptom severity. The results of this study can help clinicians identify patients who may benefit from early surgical intervention.
  Interventions: Diagnostic Test: CTQ-SSS scores

INTERVENTIONS:
Diagnostic Test: CTQ-SSS scores — The CTQ-SSS is a self-reported questionnaire that measures the severity of symptoms related to carpal tunnel syndrome, including pain, numbness, tingling, and weakness in the hand and wrist.
  Participants in this study will complete the CTQ-SSS and other functional measures that include:
  1. demographic information
  2. hand dominance
  3. Boston Carpal Tunnel Questionnaire (BCTQ)
  4. nerve conduction studies (NCS) to measure median nerve conduction velocity (NCV), distal motor latency (DML), and sensory nerve action potential (SNAP) amplitude, Compound muscle action potential (CMAP) amplitude.
  5. Hand grip strength
  Outcomes will be measured at baseline, 3 months, 6 months, and 12 months.
  The primary outcome will be progression to carpal tunnel release surgery, and logistic regression models will be used to assess the predictive value of baseline CTQ-SSS scores for this outcome, adjusted for potential confounding factors such as age, sex, and baseline symptom severity.

SUMMARY:
This study aims to determine the predictive value of baseline CTQ-SSS scores for progression to carpal tunnel release (CTR) surgery in patients with carpal tunnel syndrome (CTS). It will be a prospective cohort study involving at least 200 patients with CTS who are undergoing nonsurgical management. Participants will complete the CTQ-SSS and other functional measures at baseline, 3 months, 6 months, and 12 months, and the primary outcome will be progression to CTR surgery. Logistic regression models will be used to assess the predictive value of baseline CTQ-SSS scores for progression to CTR surgery, adjusting for potential confounding factors such as age, sex, and baseline symptom severity. The results of this study can help clinicians identify patients who may benefit from early surgical intervention.

ELIGIBILITY:
Inclusion Criteria:

* Patients with symptoms consistent with carpal tunnel syndrome, such as numbness, tingling, or pain in the hand or wrist.
* Patients with a positive nerve conduction study confirming carpal tunnel syndrome, OR patients with clinical symptoms and signs consistent with carpal tunnel syndrome if a nerve conduction study is not available or inconclusive.
* Patients who have not undergone hand or wrist surgery within the past 6 months.
* Patients who are 18 years of age or older.
* Patients who are willing and able to provide informed consent and comply with study requirements.

Exclusion Criteria:

* Patients with a history of hand or wrist surgery within the past 6 months.
* Patients with severe hand or wrist pain that would prevent completion of the outcome measures or interfere with their ability to participate in the study.
* Patients with severe cognitive impairment or language barrier that would prevent understanding of the study instructions or interfere with their ability to participate in the study.
* Patients with other neurologic or musculoskeletal disorders that could affect hand function or interfere with test completion.
* Pregnant or breastfeeding women.
* Patients who have participated in another clinical trial within the past 30 days.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: The study population will consist of patients with carpal tunnel syndrome who are undergoing nonsurgical management.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2023-07-12 (Estimated); Primary Completion 2024-11-01 (Estimated); Study Completion 2024-11-01 (Estimated)

PRIMARY OUTCOMES:
Predictive value of baseline CTQ-SSS scores for progression to carpal tunnel release (CTR) surgery. | Participants will be followed up for a 12-month period.
  To determine the predictive value of baseline CTQ-SSS scores for progression to CTR surgery in patients with carpal tunnel syndrome undergoing nonsurgical management

CONTACTS AND LOCATIONS:
Overall Officials: Amal Fawzy, Ph.d, Study Chair — Faculty of Physical Therapy, Ahram Canadian University
Locations (1):
- Outpatient clinic of faculty of physical therapy, Ahram Canadian University, Al Ḩayy Ath Thāmin, Giza Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The individual participant data (IPD) collected during this study will be available upon reasonable request. Requests for access to the data should be submitted via email to mohamed.elmeligie@acu.edu.eg. All requests will be reviewed by the study investigators to ensure that they are reasonable and consistent with the ethical principles of the study. Access to the data will be granted in compliance with applicable laws and regulations, and with appropriate safeguards to protect the privacy and confidentiality of study participants.
Supporting Information: Study Protocol, SAP, ICF
Access Criteria: via email to mohamed.elmeligie@acu.edu.eg